CLINICAL TRIAL: NCT07312981
Title: The CPH-MBD Cohort - Substudy on Dietary History
Brief Title: The CPH-MBD Cohort Dietary Substudy - Comparison of Methods for Dietary Registrations
Status: Recruiting | Type: Observational
Sponsor: University of Copenhagen (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H-25039131
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: CKD; Renal Insufficiency Chronic; CKD-MBD - Chronic Kidney Disease Mineral and Bone Disorder; Pre-dialysis
Keywords: Diet; Humans; Observational; Cohort; Phosphate/urine; Calcium/urine; Mineral bone disorder; Elderly; Calcium Balance; Phosphate Balance
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess the association between the calcium and phosphorus balance and the stage of kidney disease measured by creatinine clearence in patients with chronic kidney disease stage 4 and 5. The balance is measured a measurement between the recorded diatery intake and the urinary excretion. Additionally a comparison between image based diatery accessment and weighted records will be measured

DETAILED DESCRIPTION:
All participants will be asked to take photos of all the food and fluids they consume during 24 hours. Additionally participants will be offered to weight their food and fluid for 3 days.

ELIGIBILITY:
Inclusion Criteria:

* A glomerular filtration rate of <30 ml ml/min/1.73m2
* 18 years and above

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic kidney disease stage 4-5
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2029-05-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of diatery photograph method with weighted records. | 3 days
  The intake of calcium and phosphate assesed by the 24 hour photos and the 72 hour weighing of food and fluid items will be compared.
Calcium and phosphate balance in relation to the stage of kidney disease | 3 days
  Measured by the diatery intake of calcium and phosphate in relation to the urinary calcium and phosphate excretion

SECONDARY OUTCOMES:
Urinary Calcium | 3 days
  mmol/day
Urinary phosphate | 3 days
  mmol/day
Calcium intake total and the distribution of vegetarian and animal sources | 3 days
  mg/day
Phosphate intake total and the distribution of vegetarian and animal sources | 3 days
  mg/day
sodium intake total and the distribution of vegetarian and animal sources | 3 days
  mg/day
Energy intake | 3 days
  Kcal/day
Protein intake | 3 days
  g/day
Fat intake | 3 days
  g/day
Fluid intake | 3 days
  ml/day
Plasma phosphate | 3 days
  mmol/l
Plasma calcium | 3 days
  mmol/l
Urinary creatinine | 3 days
  mmol/day
Urinary urea | 3 days
  mmol/day
Urinary sodium | 3 days
  mmol/day
Plasma FGF23 | 3 days
  mmol/l
P-calcium P- phosphate product | 3 days
  Can be calculated by multiplying plasma calcium and plasma phosphate
plasma 25-OH-Vitamin D | 3 days
  nmol/l
plasma PTH | 3 days
  pmol/l
Plasma Albumin | 3 days
  g/dl
eGFR | 3 days
  ml/min/1.73m2

CONTACTS AND LOCATIONS:
Overall Officials: Jens Rikardt Andersen, MD, MPA, Assoc Prof, Principal Investigator — University of Copenhagen
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital - Herlev, Herlev, Capital Region
  - Herlev Hospital, Dept Nephrology, Herlev

IPD SHARING:
Plan to Share IPD: No
Currently no plans for sharing